CLINICAL TRIAL: NCT02799004
Title: Opioid Prescription for Patient With Acute Pain After Discharge From Emergency Department: Ideal Duration for Adequate Relief, Adverse Events, and Addiction
Brief Title: How Much Opioids Do You Need After Your Emergency Department Visit
Status: Completed | Type: Observational
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Raoul Daoust, Researcher and Associate Professor, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Other Study IDs: 2016-1271
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients in acute pain

SUMMARY:
Pain is one of the most common complaints in emergency department (ED) and is still often poorly managed. A major prospective multicenter study reported that 74% of patients that had a pain complaint at ED triage are discharged in moderate to severe pain. Accordingly, physicians frequently prescribed analgesic after discharged for these patients, and opioid is given in 29% of ED visits involving pain complaints. However, few studies evaluate pain management after ED discharge: the frequency and length of opioids prescriptions, the opioids quantity taken by the patients, are the patients relieved and satisfied by these pain treatments, what are the adverse effects associated with the use of these medications, and what are the chances of developing addiction?

The primary aim of this study is to determine the required minimal opioids prescription for patients treated for acute pain after being discharge from the ED. Secondary objectives include: 1) monitor the patients' adverse events during opioids treatment; 2) evaluate the patients' level of pain relief associated with their respective opioids treatment; 3) determine the patients' level of addiction following post-ED opioids treatments.

The design of the project is a prospective observational cohort study. A cohort of consecutive ED patients aged 18 or more with an initial pain at triage of 4 or more and discharged from the ED in less than 48 hours with a prescription of opioid will be asked to participate in the study. Patients will be excluded if there is ongoing treatment for a pre-existing chronic pain condition or if they used opioid drugs in the past year. Research nurses will contact the patients by phone at three follow-up time points (1 week, 1 month, and 3 months). Follow-up phone interviews will evaluate pain intensity as well as pain treatment satisfaction (0-10 NRS), monitor adverse events, and investigate possible opioids addiction (SOWS: subjective opioid withdrawal scale). During these interviews, the nurses will also question the patients about their daily opioids usage and if they were relieved from pain.

This study will provide the base for future guidelines regarding the prescription of opioids treatment for specific pathology encountered in ED. It will also give indications on how to adjust the treatments according to adverse events and the level of addiction experienced by patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Pain level at 4 or greater at triage
* Acute pain (2 weeks or less)
* Opioids prescription at discharge

Exclusion Criteria:

* Language barrier
* Pregnancy
* Treated for chronic pain
* Hospital stay greater than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of consecutive emergency department patients aged 18 or more treated for an acute pain diagnosis present for less than two weeks, with an initial pain at triage of 4 and more on a 0-10 points NRS and discharged with a prescription of opioids.
  The study will take place in an emergency department of a tertiary (trauma specialized center) academic urban hospital with an annual census of approximately 60,000 ED visits.
Sampling Method: Non-Probability Sample
Enrollment: 761 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Opioids consumption | 2 weeks
  The number of opioids taken after ED discharge for a given pathology

SECONDARY OUTCOMES:
Side effects | 2 weeks
  Recorded undesirable side effect associated with post-emergency opioids treatment
Pain relief | 2 weeks
  Patients' pain relief associated with a given prescription for a specific pathology
Addiction | 3 months
  Patients opioids addiction at three month following a post-emergency prescription

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Daoust, MD MSc, Principal Investigator — Université de Montréal
Locations (1):
- Hopital du Sacre-Coeur de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daoust R, Paquet J, Cournoyer A, Piette E, Morris J, Lessard J, Lavigne G, Chauny JM. Relationship between acute pain trajectories after an emergency department visit and chronic pain: a Canadian prospective cohort study. BMJ Open. 2020 Dec 7;10(12):e040390. doi: 10.1136/bmjopen-2020-040390. PMID 33293313
- [Derived] Daoust R, Paquet J, Gosselin S, Lavigne G, Cournoyer A, Piette E, Morris J, Castonguay V, Lessard J, Chauny JM. Opioid Use and Misuse Three Months After Emergency Department Visit for Acute Pain. Acad Emerg Med. 2019 Aug;26(8):847-855. doi: 10.1111/acem.13628. Epub 2019 Jul 18. PMID 31317619
- [Derived] Daoust R, Paquet J, Cournoyer A, Piette E, Morris J, Lessard J, Castonguay V, Williamson D, Chauny JM. Side effects from opioids used for acute pain after emergency department discharge. Am J Emerg Med. 2020 Apr;38(4):695-701. doi: 10.1016/j.ajem.2019.06.001. Epub 2019 Jun 3. PMID 31182367
- [Derived] Daoust R, Paquet J, Cournoyer A, Piette E, Morris J, Lessard J, Castonguay V, Lavigne G, Chauny JM. Acute Pain Resolution After an Emergency Department Visit: A 14-Day Trajectory Analysis. Ann Emerg Med. 2019 Aug;74(2):224-232. doi: 10.1016/j.annemergmed.2019.01.019. Epub 2019 Feb 21. PMID 30797575
- [Derived] Daoust R, Paquet J, Cournoyer A, Piette E, Morris J, Gosselin S, Emond M, Lavigne G, Lee J, Chauny JM. Quantity of opioids consumed following an emergency department visit for acute pain: a Canadian prospective cohort study. BMJ Open. 2018 Sep 17;8(9):e022649. doi: 10.1136/bmjopen-2018-022649. PMID 30224393